CLINICAL TRIAL: NCT02153775
Title: Preliminary Study of Effects of Progressive Muscle Relaxation on Cigarette Craving and Withdrawal Symptoms of Experienced Smokers in Acute Cigarette Abstinence : A Randomised Control Trial
Brief Title: Progressive Muscle Relaxation and Cigarette Craving
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Rasmon Kalayasiri, Assistant Professor, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB031/55
Record Dates: First submitted 2014-05-26; First posted 2014-06-03 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-05

CONDITIONS: Addiction
Keywords: Progressive muscle relaxation; Cigarette; Smoking; Craving
MeSH Terms: conditions — Behavior, Addictive; Smoking | interventions — Autogenic Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Progressive muscle relaxation (Experimental): Progressive muscle relaxation: single 20-minutes session
  Interventions: Behavioral: Progressive Muscle Relaxation
- Reading newspaper of the day (No Intervention): Reading newspaper of the day : single 20-minutes session

INTERVENTIONS:
Behavioral: Progressive Muscle Relaxation — Comparison of progressive muscle relaxation and no intervention (e.g., reading newspaper of the day) for the same amount of time.
  Arms: Progressive muscle relaxation

SUMMARY:
Cigarette craving usually occurs with unpleasant feelings, including stress. Progressive Muscle Relaxation (PMR) may reduce level of cigarette craving and/or withdrawal symptoms.

DETAILED DESCRIPTION:
The study reports on a study investigating the acute effects of a one-time application of progressive muscle relaxation on craving for cigarettes in smokers who were instructed to abstain from cigarettes for 3 hours.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or more
* Daily cigarette smokers

Exclusion Criteria:

* Hospitalization
* Participating in cigarette dependency treatment or trying to quit smoking with other methods
* Uncontrolled blood pressure
* Current other substance users (except alcohol)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Craving | Immediately after a 20-minutes session of progressive muscle relaxation
  Craving, a strong desire for using a substance when abstaining from substance, was measured by the Penn Alcohol Rating Scale - adapted (PACS-adapted) and the Visual Analog Scale (VAS).

SECONDARY OUTCOMES:
Cigarette withdrawal-related and non-withdrawal related feelings | Immediately after a 20-minutes session of progressive muscle relaxation
  Cigarette withdrawal symptoms (i.e., anxious, hungry, feeling bad, restless) and non-withdrawal (i.e., high, stimulated, paranoid, tongue - tied) (59-61), as measured by using the Visual Analog Scale (VAS)

OTHER OUTCOMES:
Blood pressure | Immediately after a 20-minutes session of progressive muscle relaxation
  Systolic and diastolic blood pressure, measured by an automated machine
Pulse rate | Immediately after a 20-minutes session of progressive muscle relaxation
  Pulse rate, measured by an automated machine

CONTACTS AND LOCATIONS:
Overall Officials: Thatsanee Limsanon, M.Sc., Principal Investigator — Chulalongkorn University
Locations (1):
- Department of Psychiatry, Faculty of Medicine, Chulalongkorn University, Bangkok, Bangkok, Thailand

REFERENCES:
- [Derived] Limsanon T, Kalayasiri R. Preliminary effects of progressive muscle relaxation on cigarette craving and withdrawal symptoms in experienced smokers in acute cigarette abstinence: a randomized controlled trial. Behav Ther. 2015 Mar;46(2):166-76. doi: 10.1016/j.beth.2014.10.002. Epub 2014 Nov 7. PMID 25645166
- See also: Thesis description — http://thesis.grad.chula.ac.th/current.php?mode=show&id=5474122930